CLINICAL TRIAL: NCT07198620
Title: Efficacy and Safety of IBI351 in Chinese Patients With KRAS G12C-Mutant Advanced NSCLC: A Retrospective Real-World Study
Brief Title: A Real-World Study of IBI351 for KRAS G12C+ NSCLC in China
Status: Not yet recruiting | Type: Observational
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Sponsor
Other Study IDs: CTONG2507
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-08

CONDITIONS: Lung Cancer (NSCLC)
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- IBI351 treatment: Patients with KRAS G12C-Mutant Advanced NSCLC Treated with IBI351

SUMMARY:
This study is a retrospective, multicenter, real-world investigation designed to evaluate the efficacy and safety of IBI-351 in Chinese patients with advanced non-small cell lung cancer (NSCLC) harboring a KRAS G12C mutation in a real-world setting. A total of 600 patients with KRAS G12C-mutated advanced NSCLC who received treatment with IBI-351 between August 2024 and August 2025 will be retrospectively enrolled. Descriptive statistical methods will be used to summarize the baseline characteristics, demographic data, and medication profiles of the subjects. Unless otherwise specified, continuous data will be described using counts, means, standard deviations, maximum and minimum values, and medians; categorical data will be summarized using counts and percentages. The incidence of adverse events (AEs) and serious adverse events (SAEs) will be aggregated and presented as the number and percentage of affected subjects, and all AEs will be listed in detail. The primary endpoint is the objective response rate (ORR) as assessed by investigators, and descriptive statistics for ORR will be provided. For the secondary endpoints, progression-free survival (PFS) and overall survival (OS), Kaplan-Meier (K-M) analysis will be performed to estimate median values and corresponding 95% confidence intervals (CIs), and K-M curves will be generated accordingly.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily participate in the study and provide signed informed consent.
* Have histologically or cytologically confirmed locally advanced or metastatic NSCLC, classified according to the IASLC 8th edition Lung Cancer TNM Staging System.
* Carry a confirmed KRAS G12C mutation via molecular testing.
* Have received at least one dose of oral IBI-351 treatment between August 2024 and August 2025.

Exclusion Criteria:

* Histologically or cytologically confirmed mixed NSCLC with a predominant small cell or squamous cell carcinoma component.
* Presence of EGFR sensitizing mutations, ALK rearrangements, ROS1 fusions, or other genomic alterations for which NMPA has approved first-line NSCLC therapies.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with KRAS G12C-Mutant Advanced NSCLC Treated with IBI351
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | At least 12 months retrospectively
  The proportion of patients achieving complete and partial response after treatment, measured according to RECIST v1.1 criteria

SECONDARY OUTCOMES:
Time to treatment discontinuation | At least 12 months retrospectively
  The time from the initiation of IBI351 to the patient discontinuing the medication for any reason
Progression-free survival | At least 12 months retrospectively
  defined as the time from first dose of IBI351 to the first documentation of disease progression or death from any cause, whichever occurs first. Disease progression will be assessed according to RECIST version 1.1 criteria.
Overall survival | At least 12 months retrospectively
  The time from the first administration of IBI351 to death due to any reason
Adverse events | At least 12 months retrospectively
  Assessed by recording treatment-related adverse events and serious adverse events , graded according to the CTCAE version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong Provincial People's Hospital, Guangdong Academy of Medical Sciences, Southern Medical University,, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided